CLINICAL TRIAL: NCT05288972
Title: The Effect of Different Mattress Types on Sleep Quality, Pain, Fatigue, Physical Adaptation, Functional Status, and Quality of Life in Adult Individuals With Idiopathic Scoliosis
Brief Title: The Effect of Different Mattress Types on Sleep Quality in Adult Individuals With Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Yataş Yatak ve Yorgan San. Tic. A.Ş. (Unknown)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Asst.Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: gGqs42M4
Record Dates: First submitted 2022-03-07; First posted 2022-03-21 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Idiopathic Scoliosis; Sleep
Keywords: spine; scoliosis; mattress; fatique; pain; quality of life
MeSH Terms: conditions — Scoliosis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mattress 1 (Experimental): Mattress 1 group will receive Polyurethane, Bonnel spring, medium-hard mattress
  Interventions: Device: Mattress 1
- Mattress 2 (Active Comparator): Mattress 2 group will receive Polyurethane, pocket spring, medium mattress
  Interventions: Device: Mattress 2

INTERVENTIONS:
Device: Mattress 1 — A mattress (M1) with the technical features suitable for scoliosis with supports the spine properly. The mattress will use for 4 weeks, at least 5 days a week, including at least 6 hours of sleep per day.
  Arms: Mattress 1
Device: Mattress 2 — A mattress with standard technical features (M2). The mattress will use for 4 weeks, at least 5 days a week, including at least 6 hours of sleep per day.
  Arms: Mattress 2

SUMMARY:
Objective: The aim of this study is to investigate the effect of different mattress materials on sleep behavior in adults with idiopathic scoliosis treated with non-invasive techniques.

Hypothesis 0: The use of a mattress that supports the spine properly, together with sleep accessories such as pillows, does not affect sleep behavior, does not alleviate back pain, and does not affect overall sleep quality and duration in adults with scoliosis.

Hypothesis 1: The use of a mattress that supports the spine properly, along with sleep accessories such as pillows, affects sleep behavior, helps relieve back pain, and affects overall sleep quality and duration in adults with scoliosis.

Possible outcomes: Improving sleep behavior and supporting the quality of life of individuals with idiopathic scoliosis.

DETAILED DESCRIPTION:
Scoliosis, which is characterized by the curvature of the spine to the right or left, is a common orthopedic problem today. Due to the restriction of mobility and various symptoms of the disease, people may experience difficulties in their daily lives. The clinical manifestation of scoliosis in adults is most often characterized by the presence of back pain. Unbalanced, overloaded, and strained back muscles are under constant pressure and contribute greatly to back pain. The pain may be localized at the apex of the curve (apex) or around the concavity or may radiate down the leg. This can affect people's fatigue, physical adaptation, functional status, and quality of life. This study aims to examine sleep behavior and to investigate the effects of different mattress materials on pain, sleep quality, fatigue, physical adaptation, functional status, and quality of life in adults with idiopathic scoliosis treated with non-invasive techniques.

Voluntary participants who have been diagnosed with idiopathic scoliosis will be included in the study. Signed voluntary consent will be obtained from participants. The participants will be divided into 2 groups by block randomization according to the curve type and severity and will be evaluated as double-blind.

The first group will be given a mattress (M1) with the technical features suitable for scoliosis with supports the spine properly, and the control group will be given a mattress with standard technical features (M2). The mattresses will use for 4 weeks, at least 5 days a week, including at least 6 hours of sleep per day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic scoliosis
* Cobb angle between 10 and 50 degrees
* Age 18-45 years
* Last mattress use period > 6 months

Exclusion Criteria:

* Surgical history (last 2 years)
* Lung problems, chronic respiratory or neuromuscular disease,
* Back Depression Scale score ≥ 17 & taking antidepressants
* Insomnia Severity Index score ≥ 7 & Using sleeping pills/hormones
* Diagnosed with a sleep disorder (history of restless sleep, sleep apnea…)
* Non-vertebral pain that affects sleep behavior
* Presence of a newly developed condition in the last 6 months that will affect sleep quality
* A change in the conservative treatment for scoliosis in the last 3 months, or a change is planned
* BMI <18.5 or >30 kg/m2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-03 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Self Reported Sleep Quality | 4 weeks
  Pittsburgh Sleep Quality Scale: It is a 19-item self-report scale that evaluates sleep quality and disturbance in the past month. Each item of the test is scored equally between 0-3. The scale consists of 7 subscales that assess subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleep medication, and loss of daytime functionality. By summing up the subscales, a total score ranging from 0 to 21 is obtained. A total score greater than five, with 89.6% sensitivity and 86.5% specificity, indicates inadequate sleep quality and indicates severe impairment in at least two of the above-mentioned areas or moderate impairment in three areas.
Sleep Quality with Wearable Actigraph | 1 week
  Wearable Actigraph: The wearable actigraphs to be used in the study are small, lightweight, portable devices that can be worn in the form of a watch, measuring sleep and wake cycles, and sensitively detecting motor activities.
  In the study, wearable sleep actigraphs (Actigraph wgt3x-bt) will be used by attaching them to the non-dominant wrists of the participants, thus enabling the recording and storage of resting and activity patterns in a digital environment. Each participant will be asked to wear the wearable sleep actigraph in the form of a watch for 7 days (5 weekdays and 2 weekend days) during the last week of the study, and sleep data will be recorded. The recorded data will be transferred to the computer and after the transfer, the device will be reformatted and prepared for new recordings.
Sleep Quality with Non-Wearable Actigraph | 4 weeks
  Non-Wearable Actigraph: Non-wear actigraphs (Reston Z200) to be used in the study are made ready for use by laying them on the bed. While the cord of the device is laid inside the bed, the device is suspended from the side of the bed. Bed linen is placed on it. Thus, it does not disturb the person during sleep. Each participant will be asked to use the no-wear sleep actigraph laid on their bed every day (5 weekdays and 2 weekend days) throughout the study (4 weeks). With a free application installed on the smartphone, 30 days of sleep data will be recorded.

SECONDARY OUTCOMES:
Subjective Feedback Inquiry | 4 weeks
  Subjective Feedback Questionnaire: It consists of questions such as the feeling of comfort in nine body regions (neck, shoulder, back, elbows, waist, hand/wrist, hip/thigh, knee, ankle), feeling of firmness, preference for bed, preference for sinking-buried. It will be marked on a 5-point Likert scale. Scoring is done between 0-5 for each. The higher the score represents better comfort.
Pain intensity | 4 weeks
  Visual Analog Scale (VAS): Patients will be asked to mark the degree of pain they feel at rest, in motion, and at night on the 10 cm VAS line. The condition that there is no pain is expressed as 0, and the condition that there is too much pain to be tolerated is expressed as 10. Subjects are asked to rate the pain they feel in their back/waist in the evening (before going to bed), at night (sleeping), in the morning (when getting out of bed in the morning), during the day (during the day). High scores indicate an increasing degree of pain.
Musculoskeletal Discomfort | 4 weeks
  Cornell Musculoskeletal Questionnaire (CMQ): It's a 54-item questionnaire and involves a self-rating of the frequency, severity, and work interference of the musculoskeletal discomfort on three scales across 20 body parts. On the frequency scale, the frequency of experiencing musculoskeletal discomfort in the past week is rated as never(0), 1-2 times per week(1.5), 3-4 times per week(3.5), every day(5), several times per day(10). On the severity scale, the severity of the experienced musculoskeletal discomfort is rated across the following anchors: 'Slightly uncomfortable'(1), 'Moderately uncomfortable (2), and 'Very uncomfortable'(3). On the work interference scale, the interference of the experienced musculoskeletal discomfort with the ability to work is rated across the following anchors: 'Not at all'(1), 'Slightly interfered'(2), and 'Substantially interfered'(3). High scores signify that discomfort frequency, severity, and working ability interference are high.
Fatigue | 4 weeks
  Multidimensional Assessment of Fatigue (MAF): The scale contains 16 items and measures four dimensions of fatigue: severity (1-2), distress (3), degree of interference in activities of daily living (4-14), and timing (15-16). Scores range from 1 (no fatigue) to 50 (severe fatigue).
Functional Status | 4 weeks
  The Functional Rating Index (FRI): FRI is a self-reporting instrument consisting of 10 items, each with 5 possible responses (0-4) that express graduating degrees of disability. Scoring ranges from 0-40, and the higher the score, the worse the functional status.
Trunk Sagittal Plane Flexibility | 4 weeks
  Finger-to-floor test: Finger-to-floor distance test was used to measure lumbar mobility. This test measures the maximal possible spinal flexion range, and the participants bent their bodies forward without flexing their knees until there was a functional limitation. The distance between the tip of the right middle finger and the floor was measured as the finger-to-floor distance score (cm) using standard tape. Higher distances were indicative of greater hamstring tightness and limited lumbopelvic mobility.
Trunk Frontal Plane Flexibility | 4 weeks
  Finger-to-floor test: Finger-to-floor distance test was used to measure lumbar mobility. This test measures the maximal possible spinal flexion range, and the participants laterally flexed their bodies forward without flexing their knees until there was a functional limitation. The distance between the tip of the third digit and the floor was measured (cm) using standard tape. Higher distances were indicative of greater frontal plane lumbopelvic mobility.
Trunk Endurance | 4 weeks
  Static endurance of trunk muscles will be evaluated in plank position, supine hook lying position with the trunk flexed to 60 degrees, in the prone Biering-Sorenson Test position (prone with the upper body and abdomen off the edge of the table), and side bridge position. The ability to maintain these positions will be recorded in seconds with a chronometer. Higher time duration indicates higher muscular endurance.
The Quality of Life | 4 weeks
  The Nottingham Health Profile (NHP): It is a 38-item questionnaire that assesses the domains of physical mobility, pain, sleep, social isolation, emotional reactions, and energy level. All questions have only yes/no answer options and each section score is weighted. Its wording is simple and easily understood, and can be completed by patients in 5 minutes. High scores indicate a decrease in quality of life. The highest score in any section is 100.
Soliosis Specific Quality of Life | 4 weeks
  Scoliosis Research Society-22 Questionnaire (SRS-22): The questionnaire assesses five domains: function, pain, personal image, mental health (five questions each) and treatment satisfaction (two questions). Each question is scored between 1 (worst) and 5 (best). In the interrogation whose total score ranged from 22 to 111, the high score indicates that the quality of life for scoliosis is better.

CONTACTS AND LOCATIONS:
Overall Officials: Ipek Yeldan Karagoz, Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Faculty of Health Science, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No